CLINICAL TRIAL: NCT00652093
Title: Lumbar Stenosis Outcomes Research II: Opana IR Versus Placebo and Active Control (Darvocet) for the Treatment of Walking Impairment in Lumbar Spinal Stenosis: A Double-Blind Randomized, Cross-Over Trial
Brief Title: Lumbar Stenosis Outcomes Research II
Acronym: LUSTORII
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Removal of Darvocet from US market
Sponsor: University of Rochester (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John Markman, Director, Translational Pain Research, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20957
Record Dates: First submitted 2008-03-11; First posted 2008-04-03 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Oxymorphone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Opana then darvocet then placebo (Experimental): Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the second study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the third study visit, four days later placebo tablet was given one time at the fourth study visit.
  Interventions: Drug: opana then darvocet then placebo
- Opana then placebo then darvocet (Experimental): Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the second study visit, four days later placebo tablet was given one time at the third study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the fourth study visit.
  Interventions: Drug: opana then placebo then darvocet
- Placebo then opana then darvocet (Experimental): Placebo tablet tablet was given one time at the second study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) was given one time at the third study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the fourth study visit.
  Interventions: Drug: placebo then opana then darvocet
- Placebo then darvocet then opana (Experimental): Placebo tablet tablet was given one time at the second study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the third study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the fourth study visit.
  Interventions: Drug: Placebo then darvocet then opana
- Darvocet then opana then placebo (Experimental): Darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the second study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the third study visit, four days later placebo tablet was given one time at the fourth study visit.
  Interventions: Drug: Darvocet then opana then placebo
- Darvocet then placebo then opana (Experimental): Darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the second study visit, four days later placebo tablet was given one time at the third study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the fourth study visit.
  Interventions: Drug: Darvocet then placebo then opana

INTERVENTIONS:
Drug: opana then darvocet then placebo — Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the second study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the third study visit, four days later placebo tablet was given one time at the fourth study visit.
  Other Names: opana: oxymorphone HCL; darvocet: propoxyphene/acetaminophen; placebo: inactive drug
  Arms: Opana then darvocet then placebo
Drug: opana then placebo then darvocet — Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the second study visit, four days later placebo tablet was given one time at the third study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the fourth study visit.
  Other Names: opana: oxymorphone HCL; darvocet: propoxyphene/acetaminophen; placebo: inactive drug
  Arms: Opana then placebo then darvocet
Drug: placebo then opana then darvocet — Placebo tablet tablet was given one time at the second study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) was given one time at the third study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the fourth study visit.
  Other Names: opana: oxymorphone HCL; darvocet: propoxyphene/acetaminophen; placebo: inactive drug
  Arms: Placebo then opana then darvocet
Drug: Placebo then darvocet then opana — Placebo tablet tablet was given one time at the second study visit, four days later darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the third study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the fourth study visit.
  Other Names: opana: oxymorphone HCL; darvocet: propoxyphene/acetaminophen; placebo: inactive drug
  Arms: Placebo then darvocet then opana
Drug: Darvocet then opana then placebo — Darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the second study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the third study visit, four days later placebo tablet was given one time at the fourth study visit.
  Other Names: opana: oxymorphone HCL; darvocet: propoxyphene/acetaminophen; placebo: inactive drug
  Arms: Darvocet then opana then placebo
Drug: Darvocet then placebo then opana — Darvocet (100mg Propoxyphene/650mg Acetaminophen) tablet was given one time at the second study visit, four days later placebo tablet was given one time at the third study visit, four days later Opana IR, 5mg (oxymorphone hydrochloride) tablet was given one time at the fourth study visit.
  Other Names: opana: oxymorphone HCL; darvocet: propoxyphene/acetaminophen; placebo: inactive drug
  Arms: Darvocet then placebo then opana

SUMMARY:
The primary objective of the proposed pilot study is to determine the efficacy of oxymorphone hydrochloride and propoxyphene/acetaminophen combination in prolonging the time to onset of pain and reducing the severity of pain associated with walking in patients lumbar spinal stenosis that have clinical symptoms of neurogenic claudication. Neurogenic claudication is defined as movement induced leg pain, numbness, heaviness, or vague discomfort in part or all of one or both legs provoked with walking and standing and relieved by sitting, squatting, or forward flexion posturing. The secondary objective is to examine the functional benefit of oxymorphone hydrochloride and propoxyphene/acetaminophen combination with respect to improvement in duration and distance of walking.

DETAILED DESCRIPTION:
A computer-generated randomization plan was used for assignment of subjects to one of six treatment sequences (4 subjects per sequence): oxymorphone/propoxyphene/placebo, oxymorphone/placebo/propoxyphene, placebo/oxymorphone/propoxyphene, placebo/propoxyphene/oxymorphone, propoxyphene/oxymorphone/placebo, or propoxyphene/placebo/oxymorphone. One dose of blinded study drug (opana, propoxypehen, or placebo) was given at study days 1, 5, and 9. The primary endpoint was time to first symptoms of moderate intensity (NRS ≥ 4/10) during treadmill ambulation. Ambulation assessment was performed during the screening visit. Ambulation assessment was also performed 90 minutes after administration of study drug on days 1, 5 and 9, to evaluate pain intensity associated with walking as well as distance covered by the patients. Quantitative assessment of ambulation was conducted on a treadmill at 0° ramp incline at 1.2 miles per hour (mph). Measurement of self-reported symptom severity using the NRS at baseline, and every 30 seconds for a maximum of 15 minutes was recorded. The following information was also recorded: time to first symptoms, total ambulation time. The examination was stopped after 15 minutes or at the onset of severe symptoms. Severe symptoms were defined as the level of discomfort that would make patients stop walking in usual life situations. No one was encouraged or prompted to continue walking beyond this point. Patients were instructed to walk with an upright posture. They were not permitted to lean forward or hold onto the handrails during the examination. Secondary outcome measures included area under the curve of present pain intensity with ambulation at each specified time point, final pain intensity with walking, walking tolerance, time to return to baseline pain level after ambulation, as well as the results of a series of pain related questionnaires including: Visual Analog Scale (VAS), Patient Global Assessment (PGA), NRS, Roland Morris Disability Questionnaire (RMDQ), modified Brief Pain Inventory short form (mBPI-sf), Oswestry Disability Index (ODI), and Swiss Spinal Stenosis (SSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients must present with clinical symptoms of neurogenic claudication (exercise induced leg pain, numbness, heaviness, or vague discomfort in part or all of one or both legs provoked with walking and standing and relieved by sitting, squatting, or forward flexion posturing) and endorse limitation of walking tolerance due to these symptoms
* Numeric Rating Scale (NRS) for pain ≥ 6 in response to the following question: "Circle one number (from 0=no pain to 10=worst pain) - How would you rate the worst leg and lower back pain you experienced during walking last week?"
* Patients must have confirmatory imaging by MRI or CT scan demonstrating at least one level of lumbar spinal stenosis within 1 year
* Duration of symptoms > 3 months
* Age > 50 years; male or female

Exclusion Criteria:

* Past or present existence of a movement disorder, e.g., Parkinsonism, or an neurologic disease that might affect the ability to ambulate (e.g., signs/symptoms of cauda equina compression)
* Cognitive impairment preventing full understanding or participation in the study
* Peripheral vascular disease
* Moderate to severe arthritis of the knee or hip that might severely compromise ambulation
* Past or present lower extremity peripheral vascular disease
* Serious concomitant medical illness (e.g., heart disease) that might impair ambulation assessment
* Previous lumbar surgery for spinal stenosis (laminectomy with or without fusion) within the past 2 years or epidural steroid injection in the preceding 4 months.
* Severe psychiatric disorder
* Mean time to severe symptoms > 15 minutes.
* Epidural steroid treatment within the last three months
* History of drug or alcohol dependence
* Serious intercurrent illness
* Hypersensitivity to oxymorphone hydrochloride
* Hypersensitivity to propoxyphene or acetaminophen
* Severe bronchial asthma or hypercarbia, morphine analogs such as codeine, or any of the other ingredients of Opana
* Suspicion of paralytic ileus
* Moderate or severe hepatic impairment
* Major conduction abnormality on ECG or cardiac (Bruce protocol) stress test within the past year.
* Ongoing treatment with a long-acting opioid or regularly-scheduled use of a short acting opioid (>3 doses/day on four or more days/week).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Markman, M.D., Principal Investigator — University of Rochester
Locations (1):
- 2180 S. Clinton Ave, Rochester, New York, United States

REFERENCES:
- [Background] Simon LS, Evans C, Katz N, Bombardier C, West C, Robbins J, Copley-Merriman C, Markman J, Coombs JH. Preliminary development of a responder index for chronic low back pain. J Rheumatol. 2007 Jun;34(6):1386-91. PMID 17552065
- [Background] Markman JD, Dworkin RH. Ion channel targets and treatment efficacy in neuropathic pain. J Pain. 2006 Jan;7(1 Suppl 1):S38-47. doi: 10.1016/j.jpain.2005.09.008. PMID 16427000
- [Background] Deen HG Jr, Zimmerman RS, Lyons MK, McPhee MC, Verheijde JL, Lemens SM. Test-retest reproducibility of the exercise treadmill examination in lumbar spinal stenosis. Mayo Clin Proc. 2000 Oct;75(10):1002-7. doi: 10.4065/75.10.1002. PMID 11040847
- [Background] Deen HG, Zimmerman RS, Lyons MK, McPhee MC, Verheijde JL, Lemens SM. Use of the exercise treadmill to measure baseline functional status and surgical outcome in patients with severe lumbar spinal stenosis. Spine (Phila Pa 1976). 1998 Jan 15;23(2):244-8. doi: 10.1097/00007632-199801150-00019. PMID 9474733
- [Background] Stucki G, Daltroy L, Liang MH, Lipson SJ, Fossel AH, Katz JN. Measurement properties of a self-administered outcome measure in lumbar spinal stenosis. Spine (Phila Pa 1976). 1996 Apr 1;21(7):796-803. doi: 10.1097/00007632-199604010-00004. PMID 8779009
- [Derived] Markman JD, Gewandter JS, Frazer ME, Murray NM, Rast SA, McDermott MP, Chowdhry AK, Tomkinson EJ, Pilcher WH, Walter KA, Dworkin RH. A Randomized, Double-blind, Placebo-Controlled Crossover Trial of Oxymorphone Hydrochloride and Propoxyphene/Acetaminophen Combination for the Treatment of Neurogenic Claudication Associated With Lumbar Spinal Stenosis. Spine (Phila Pa 1976). 2015 May 15;40(10):684-91. doi: 10.1097/BRS.0000000000000837. PMID 25705958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 08 December 2007 (initial IRB approval) to 26 August 2011* (final study results) First patient enrolled: 12 June 2008. Last patient completed: 12 October 2010
  *Study terminated on 29 November 2010 due to US Food and Drug Administration (FDA) removing active control (Darvocet) from the U.S. market.
Pre-assignment Details: Forty-three subjects signed the Research Subject Review Board (local IRB) approved consent form. Nineteen subjects failed screening and did not meet inclusion criteria. Twenty-four subjects met radiographic and treadmill criteria for neurogenic claudication and were randomized. Of these, 21 subjects completed all phases of the study
Period: Overall Study
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 2 | 4
Not Completed | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 0 | 1 | 2 | 4
  >=65 years | 4 | 4 | 3 | 4 | 3 | 2 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (4) | 73.0 (3.2) | 76.0 (12) | 70.0 (4.8) | 76.0 (15.2) | 63.3 (6.8) | 71.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 3 | 3 | 2 | 12
  Male | 4 | 3 | 1 | 1 | 1 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Time to First Symptoms (Tfirst) of Moderate Pain
Description: Using the Numeric Rating Scale (NRS) (0=no pain, 10=worst pain imaginable)the time to first symptoms (Tfirst) with a NRS score greater than or equal to 4 (moderate pain level), with treadmill ambulation was measured. Patients were excluded from the trial if there pain at rest was greater than or equal to 4/10.
Time Frame: study visit
Population: The analyses included all 24 enrolled randomized subjects based on inclusion/exclusion criteria except for three who withdrew from trial prior to completion of study. One dropped out (physician decision) due to an adverse event (AE) (dizzy) and two dropped due to scheduling. This singular AE is not included in the AE reporting below.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
minutes | 1.73 (1.68) | 3.02 (2.90) | 3.93 (3.22) | 2.65 (3.23) | 0.83 (0.73) | 5.43 (4.28)

2. Secondary Outcome: Area Under the Curve
Description: Subjects were instructed to walk on the treadmill and to tell the research coordinator to stop testing when they reached the point at which they typically would need to stop and sit down, or until 15 minutes had elapsed. At defined intervals (every 30 seconds) subjects were asked what their pain level was according to the NRS. The area under the curve of present pain intensity is the total area combined for the amount of time the subject walked.
Time Frame: study visit
Population: Outcome measures were obtained for all subjects as described in the Analysis Population Description of the primary outcome above.
Measure: Mean (Standard Deviation); unit: units on a scale * minutes
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale * minutes | 76.0 (39.5) | 95.7 (27.7) | 95.0 (35.9) | 86.4 (39.0) | 123.3 (6.3) | 79.6 (31.5)

3. Secondary Outcome: Total Distance
Description: Subjects were instructed to walk on the treadmill and to tell the research coordinator to stop testing when they reached the point at which they typically would need to stop and sit down, or until 15 minutes had elapsed. When the subject reached their maximum distance, the treadmill testing was stopped. This was recorded as total distance based on number of minutes and seconds walked. Minutes was converted to meters based on calculation of defined speed of the treadmill.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
meters | 266.6 (191.3) | 249.5 (109.4) | 177.9 (139.1) | 290.1 (176.0) | 160.8 (96.5) | 294.8 (133.2)

4. Secondary Outcome: Recovery Time
Description: After the subject completed the treadmill test they were asked to immediately return to the seated position. At this point a timer was started. When the subjects pain level returned to baseline (level of pain subject felt in a seated position before walking) the time was stopped. This was recorded as recovery time. Maximum recovery time is 15 minutes.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
minutes | 1.10 (0.98) | 1.50 (1.37) | 2.02 (2.68) | 1.58 (1.22) | 2.15 (1.18) | 1.57 (1.19)

5. Secondary Outcome: Visual Analog Scale (VAS)
Description: The VAS asked subjects to place a mark indicative of their low back pain during the past day on a 100mm line, with 0mm representing no pain and 100mm representing extreme pain.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 51.3 (22.0) | 57.9 (25.7) | 56.2 (28.6) | 46.7 (24.0) | 63.3 (31.0) | 55.1 (30.7)

6. Secondary Outcome: Patient Global Assessment (PGA)
Description: Subjects were asked to rate their low back pain according to the PGA. PGA is the impact of disease activity. PGA was measured on a 5-point scale, where 1=very good, 2=good, 3=fair, 4=poor, and 5=very poor.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 2.8 (0.6) | 2.8 (1.0) | 3.1 (1.2) | 2.6 (0.5) | 3.3 (0.5) | 2.6 (1.1)

7. Secondary Outcome: Roland Morris Disability Questionnaire (RMDQ)
Description: The RMDQ consists of 24 yes/no statements about activity limitations due to back pain. These questions center on movement, ambulation, and self-care activities. Positive (yes) answers each contribute 1 point to cumulative score with total scores ranging from 0 (no disability) to 24 (severely disabled).
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 12.8 (4.4) | 15.3 (5.0) | 13.2 (4.1) | 15.2 (2.7) | 13.7 (3.6) | 7.4 (4.3)

8. Secondary Outcome: Modified Brief Pain Inventory (mBPI)- Interference Score
Description: The mBPI is a series of questions that rates the severity and impact of pain on daily function. The questionnaire is made up of 4 pain severity items using the NRS scale, and seven 11-point pain interference scales (0 indicating no interference and 10 indicating complete interference). For the interference score, a total score of 10 indicates pain completely interferes with activities.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 3.7 (2.0) | 4.2 (1.4) | 2.7 (0.8) | 4.3 (1.3) | 6.2 (1.0) | 2.8 (2.6)

9. Secondary Outcome: Oswestry Disability Index (ODI) Score
Description: The ODI is a set of 10 questions each with five choices (maximum score of 5 points per question) designed to determine how back pain has affected the ability to manage everyday life (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and change positions). A score of 0 indicates no disability and total score of 50 would indicate 100% disability.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 37.9 (9.7) | 98.4 (5.7) | 38.0 (6.6) | 44.1 (9.7) | 37.0 (2.8) | 29.7 (13.3)

10. Secondary Outcome: Swiss Spinal Stenosis Score- Symptom Severity
Description: The SSS is a series of questions asking about symptom severity, physical function, and satisfaction. The symptom severity section is a set of 7 questions (maximum score is 5 points per question) and asks to rate pain for each question based on no pain, mild, moderate, severe or very severe pain. The total score (maximum=35) is added up and divided by seven. The maximum score for the symptom severity section (score=5) indicates very severe symptom severity.
Time Frame: study visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 2.6 (0.6) | 2.9 (0.6) | 3.2 (0.3) | 3.2 (0.7) | 3.6 (0.5) | 2.9 (0.6)

11. Secondary Outcome: Swiss Spinal Stenosis Score- Physical Function
Description: The SSS is a series of questions asking about symptom severity, physical function, and satisfaction. The physical function section is a series of 5 questions (maximum 4 points per question) and asks to rate function for each question based on comfortably, sometimes with pain, always with pain, no functional ability. The total score (max=20) is divided by five. The maximum score for the physical function section (max=4) indicates no ability to function.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 2.5 (0.4) | 2.5 (0.2) | 2.6 (0.6) | 2.6 (0.5) | 2.6 (0.2) | 2.2 (0.2)

12. Secondary Outcome: Final Pain
Description: Subjects were instructed to walk on the treadmill and to tell the research coordinator to stop testing when they reached the point at which they typically would need to stop and sit down, or until 15 minutes had elapsed. At defined intervals subjects were asked what their pain level was according to the NRS. When the subject reached their maximum distance, they were asked their NRS score. This was recorded as final pain intensity.
Time Frame: study visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 2 | 4
units on a scale | 4.6 (2.2) | 6.6 (1.6) | 6.2 (2.7) | 6.7 (2.5) | 8.0 (0.6) | 7.1 (1.9)

ADVERSE EVENTS:
Time Frame: AEs were captured for each subject from the first study visit through the final study visit (i.e. day 1 through day 9).
Arm/Group | Opana Then Darvocet Then Placebo | Opana Then Placebo Then Darvocet | Placebo Then Opana Then Darvocet | Placebo Then Darvocet Then Opana | Darvocet Then Opana Then Placebo | Darvocet Then Placebo Then Opana
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3 | 0/4 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 0/3 | 0/4 | 0/2 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opana Then Darvocet Then Placebo (N=4) | Opana Then Placebo Then Darvocet (N=4) | Placebo Then Opana Then Darvocet (N=3) | Placebo Then Darvocet Then Opana (N=4) | Darvocet Then Opana Then Placebo (N=2) | Darvocet Then Placebo Then Opana (N=4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This single adverse event occurred after darvocet administration.
Somnolence (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This single adverse event occurred after opana administration.
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — This single adverse event occurred after placebo administration.

LIMITATIONS AND CAVEATS:
This study terminated early (leading to small number of subjects analyzed) due to US Food and Drug Administration (FDA) removing active control (Darvocet) from the U.S. market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No